CLINICAL TRIAL: NCT07257016
Title: High-Flow Oxygen Therapy Via Tracheal Intubation in Neurocritical Patients
Brief Title: HFTO Via Tracheal Intubation in Neurocritical Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Chen Guangqiang, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HX-B-2025-016
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: High Flow Oxygen Therapy; Neuro ICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFTO (Experimental): Patients with delayed extubation receiving high-flow tracheal oxygen therapy.
  Interventions: Device: HFTO
- PSV (Active Comparator): Patients with delayed extubation receiving low-level pressure support ventilation.
  Interventions: Device: PSV

INTERVENTIONS:
Device: HFTO — Use a high-flow oxygen therapy system connected to the endotracheal tube via a dedicated adapter. Initial settings: Flow rate 40 L/min, FiO₂ titrated to maintain patient SpO₂ ≥ 95%.
  Arms: HFTO
Device: PSV — Continue low-level pressure support ventilation using a mechanical ventilator. Parameter settings: Pressure support (PS) 5-8 cmH₂O, PEEP 5 cmH₂O, FiO₂ ≤ 0.40.
  Arms: PSV

SUMMARY:
Neurocritical patients often require prolonged invasive ventilation due to impaired respiratory drive and airway protection deficits. While early weaning reduces complications and costs, these patients frequently pass spontaneous breathing trials (SBT) yet remain intubated solely for airway protection.

Current practice maintains low-level pressure support ventilation (5-8 cmH₂O) to offset endotracheal tube resistance. However, prolonged ventilation increases risks of ventilator-associated pneumonia (VAP) and diaphragm dysfunction. Emerging evidence suggests appropriately sized tubes may not substantially increase work of breathing (WOB).

High-flow oxygen therapy (HFOT) delivers heated, humidified oxygen at high flow rates, reducing WOB and improving oxygenation and comfort. While validated for tracheostomized patients, HFOT via tracheal intubation (HFOT-TI) remains unstudied in neurocritical populations during early weaning.

This study aims to evaluate the safety and feasibility of HFOT-TI in neurocritical patients who have passed SBT but require ongoing airway protection.

DETAILED DESCRIPTION:
Neurocritical patients, including those with traumatic brain injury, stroke, or intracranial hemorrhage, often require prolonged mechanical ventilation due to impaired respiratory drive or airway protection needs. Weaning these patients from invasive ventilation involves two key stages: liberation from mechanical support and extubation. Early weaning reduces complications, accelerates recovery, and lowers healthcare costs. Clinical guidelines advocate early weaning assessments for patients ventilated for over 24 hours, followed by spontaneous breathing trials (SBT) to confirm readiness for independent breathing. While patients passing SBT are typically extubated promptly, neurocritical patients often face delayed extubation due to impaired consciousness or inadequate airway protection, despite adequate respiratory function. In these cases, the tracheal tube primarily ensures airway protection rather than ventilatory support.

Traditionally, low-level ventilatory support (e.g., pressure support of 5-8 cmH₂O) is used to counter the inspiratory resistance of the tracheal tube and provide humidified gas. However, prolonged ventilation, even at minimal levels, may increase risks such as ventilator-associated pneumonia and diaphragm dysfunction. Evidence indicates that appropriately sized tracheal tubes may not substantially increase the work of breathing (WOB), and some patients can compensate for this resistance without ventilatory support.

High-flow oxygen therapy (HFOT), delivered via nasal cannula or tracheostomy, provides heated, humidified oxygen at high flow rates, enhancing oxygenation, reducing WOB, and improving patient comfort. Emerging evidence supports its role in facilitating weaning in tracheostomized patients and during SBT in intubated patients. However, the safety and feasibility of HFOT via tracheal intubation (HFOT-TI) in neurocritical patients during early weaning remain largely unexplored. Given the prolonged airway protection needs in this population, HFOT-TI may serve as an effective bridge to extubation, potentially minimizing prolonged ventilatory support and associated complications.

Investigators aimed to evaluate the safety and feasibility of HFOT-TI in neurocritical patients who have passed SBT but require ongoing airway protection. Investigators assessed changes in respiratory parameters and safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Post-neurosurgical or brain injury patients with stable intracranial status (Glasgow Coma Scale ≥ 9, Richmond Agitation-Sedation Scale score -2 to +1).
* Successful completion of a 30-minute T-piece spontaneous breathing trial (per standard SBT failure criteria).
* Poor airway protection capacity (STAGE score < 6) necessitates ongoing intubation for respiratory support, as determined by the attending physician.
* Signed informed consent (by patient or legal representative).

Exclusion Criteria:

* Contraindications to esophageal pressure monitoring (e.g., esophageal varices, recent esophageal surgery).
* History of chronic respiratory diseases (e.g., COPD, severe asthma).
* Chronic heart failure (NYHA class III-IV) or severe arrhythmia.
* Body Mass Index (BMI) > 30 kg/m².
* Pregnancy.
* Anticipated need for tracheostomy without extubation attempt
* Withdrawal of life-sustaining treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
PTPes | 48 hours
  PTPes is defined as the area enclosed by the Pcw and Pes curves during the inspiratory phase, multiplied by the respiratory rate.

SECONDARY OUTCOMES:
Pmus | 48 hours
  Pmus is defined as the maximum difference between the chest wall recoil pressure (Pcw) and the esophageal pressure (Pes) during inspiration.
ΔPes | 48 hours
  The change in Pes (ΔPes) is the difference between the Pes at the start of inspiration and the maximum negative deflection of Pes during inspiration.
Ventilator-Free Days | 28 days
  Ventilator-Free Days during the first 28 days

IPD SHARING:
Plan to Share IPD: Yes
through clinical trials
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Girard TD, Alhazzani W, Kress JP, Ouellette DR, Schmidt GA, Truwit JD, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Morris PE; ATS/CHEST Ad Hoc Committee on Liberation from Mechanical Ventilation in Adults. An Official American Thoracic Society/American College of Chest Physicians Clinical Practice Guideline: Liberation from Mechanical Ventilation in Critically Ill Adults. Rehabilitation Protocols, Ventilator Liberation Protocols, and Cuff Leak Tests. Am J Respir Crit Care Med. 2017 Jan 1;195(1):120-133. doi: 10.1164/rccm.201610-2075ST. PMID 27762595
- [Background] Janssen ML, Weller D, Endeman H, Heunks LM, Wils EJ. Physiological Effects of High-Flow Tracheal Oxygen in Tracheostomized Patients Weaning From Mechanical Ventilation. Respir Care. 2024 Sep 26;69(10):1336-1344. doi: 10.4187/respcare.11755. PMID 38772682